CLINICAL TRIAL: NCT01051856
Title: A Multicenter Mayo-initiated Randomized Controlled Trial Comparing Pancreatic Leaks After TissueLink vs SEAMGUARD After Distal Pancreatectomy (PLATS)
Brief Title: TissueLink Versus SEAMGUARD After Distal Pancreatectomy
Acronym: PLATS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The trial closed early due to poor accrual.
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 09-000362
Record Dates: First submitted 2010-01-15; First posted 2010-01-20 (Estimated); Results first posted 2015-06-12 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Distal Pancreatectomy
MeSH Terms: interventions — Radiofrequency Ablation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SEAMGUARD with bioabsorbable staple (Active Comparator): In this arm pancreatic transection will be executed using an endoscopic linear stapling device. The individual staple depth can be chosen by the operating surgeon. Bioabsorbable Mesh sleeves specifically manufactured for the chosen staple depth and cartridge length will be placed over the stapler before firing.
  Interventions: Device: SEAMGUARD with bioabsorbable staple
- TissueLink with radiofrequency ablation (Active Comparator): After pancreatic transection, with any method chosen by the operating surgeon, the pancreatic remnant will be treated with TissueLink alone for an ablation depth (thickness) of approximately 7 mm using electrosurgical generator settings of 100 W and a saline drip rate of 1-2 drops per second.
  Interventions: Procedure: TissueLink with radiofrequency ablation

INTERVENTIONS:
Device: SEAMGUARD with bioabsorbable staple — In the SEAMGUARD group, pancreatic resection and transection of the pancreatic body will be executed using an endoscopic linear stapling device.
  Arms: SEAMGUARD with bioabsorbable staple
Procedure: TissueLink with radiofrequency ablation — After pancreatic transection with the method of choice of the operating surgeon, the pancreatic remnant will be treated with Tissuelink alone for an ablation depth (thickness) of approximately 7 mm.
  Arms: TissueLink with radiofrequency ablation

SUMMARY:
The purpose of this research study is to find a lowest leak rate following a distal pancreatectomy (removal of the left side of the pancreas). Distal pancreatectomy is known to have a risk of pancreatic leaks (leakage of pancreatic fluid from the cut surface of the pancreas). Two FDA cleared devices (TissueLink and SEAMGUARD) will be studied to treat and prevent leaks at the end of the pancreas.

DETAILED DESCRIPTION:
The objective of this trial is to compare the effectiveness of TissueLink closure of pancreatic stump after distal pancreatectomy to that of SEAMGUARD reinforced stapler closure.

Distal pancreatectomy is performed for a broad variety of indications including benign and malignant conditions. Specifically, distal pancreatectomy refers to resection of the portion of pancreas to the left of the superior mesenteric vein/portal vein trunk, excluding the duodenum and distal bile duct. Pancreatic duct leak at the resection margin is one of the most common complications of distal pancreatectomy. This complication prolongs in-patient and outpatient care and resulting in significant detriments to the patient's operative experience and increases in the financial burden of pancreatic surgery.

ELIGIBILITY:
Inclusion criteria:

1. Age equal or above 18 years
2. Accepted for elective distal pancreatectomy for any indication

Exclusion from randomization process:

* Thickness of pancreas on preoperative CT scan images > 2.5 cm at the site of expected transection in anterior-posterior diameter. This will be reviewed by the surgeon the day before the surgeon sees the patient to predetermine the appropriateness of the patient for the study.

General study exclusion criteria:

1. Current immunosuppressive therapy
2. Chemotherapy within 2 weeks before operation
3. Bevacizumab (Avastin™) treatment not completed at least 6 weeks before operation
4. Radiotherapy before operation
5. Inability to follow the instructions given by the investigator
6. Lack of compliance
7. Persons unable or unwilling to give informed consent to participate in this study
8. Pregnant women
9. Prisoners
10. Institutionalized individuals

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2009-12; Primary Completion 2014-03 (Actual); Study Completion 2015-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Florencia G Que, M.D. S, Principal Investigator — Mayo Clinic, Rochester, MN
Locations (2):
- United States (2):
  - Massachusettes General Hospital, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota

REFERENCES:
- [Background] Bassi C, Dervenis C, Butturini G, Fingerhut A, Yeo C, Izbicki J, Neoptolemos J, Sarr M, Traverso W, Buchler M; International Study Group on Pancreatic Fistula Definition. Postoperative pancreatic fistula: an international study group (ISGPF) definition. Surgery. 2005 Jul;138(1):8-13. doi: 10.1016/j.surg.2005.05.001. PMID 16003309
- [Derived] Shubert CR, Ferrone CR, Fernandez-Del Castillo C, Kendrick ML, Farnell MB, Smoot RL, Truty MJ, Que FG. A multicenter randomized controlled trial comparing pancreatic leaks after TissueLink versus SEAMGUARD after distal pancreatectomy (PLATS) NCT01051856. J Surg Res. 2016 Nov;206(1):32-40. doi: 10.1016/j.jss.2016.06.034. Epub 2016 Jun 17. PMID 27916372

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled from January 2010 to March 2014 at Mayo Clinic in Rochester, Minnesota, and at Massachusetts General Hospital in Boston, Massachusetts.
Period: Overall Study
Arm/Group | SEAMGUARD With Bioabsorbable Staple | TissueLink With Radiofrequency Ablation
Started | 33 | 35
Completed | 32 | 35
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SEAMGUARD With Bioabsorbable Staple | TissueLink With Radiofrequency Ablation | Total
Number analyzed (Participants) | 32 | 35 | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.84 (12.73) | 56.29 (12.79) | 57.99 (12.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 23 | 39
  Male | 16 | 12 | 28
Region of Enrollment [Number; unit: participants]
  United States | 32 | 35 | 67
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — 34 participants in the TissueLink arm were included in the BMI analysis; the data were not available on one participant.
  kg/m^2 | 27.60 (5.08) | 28.56 (5.25) | 28.09 (5.15)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Developed a Postoperative Pancreatic Duct Leak at the Resection Margin (Pancreatic Fistula) Within 90 Days From the Operation
Description: Pancreatic fistula was defined as amylase-rich (greater than 3 times upper limit of normal serum amylase for the treating institution) fluid either in the operatively placed drain or upon reinsertion of an image-guided drain for postoperative fluid collection.
Time Frame: 90 days from the operation
Population: Intention-to-treat analysis
Measure: Number; unit: percentage of subjects
Arm/Group | SEAMGUARD With Bioabsorbable Staple | TissueLink With Radiofrequency Ablation
Number analyzed (Participants) | 32 | 35
percentage of subjects | 12.5 | 22.9
Statistical Analysis 1: Comparison: SEAMGUARD With Bioabsorbable Staple vs TissueLink With Radiofrequency Ablation; Test type: Superiority or Other; p = 0.35, Chi-squared

2. Secondary Outcome: Severity of the Pancreatic Fistula Leaks
Description: Grading of the clinical severity of the leak was done according to the International Study Group on Pancreatic Fistula criteria. Severity of fistula was reported as clinically significant (Grades B and C) or not (Grade A). Grade C indicates the most severe clinical outcome.
Time Frame: 90 days post operative
Measure: Number; unit: Pancreatic fistula leaks
Arm/Group | SEAMGUARD With Bioabsorbable Staple | TissueLink With Radiofrequency Ablation
Number analyzed (Participants) | 32 | 35
Pancreatic fistula leaks
  Clinically significant pancreatic fistula leaks | 4 | 8
  Non-clinically significant pancreatic fistula leak | 11 | 14

ADVERSE EVENTS:
Time Frame: Adverse events were collected within the 90 day perioperative period.
Arm/Group | SEAMGUARD With Bioabsorbable Staple | TissueLink With Radiofrequency Ablation
Serious Adverse Events (participants affected / at risk) | 4/32 | 5/35
Other Adverse Events (participants affected / at risk) | 15/32 | 23/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEAMGUARD With Bioabsorbable Staple (N=32) | TissueLink With Radiofrequency Ablation (N=35)
Hospital readmission for pancreatic fistula (Gastrointestinal disorders) | 4 (4) | 5 (5)
Percutaneous Drainage (Surgical and medical procedures) | 4 (4) | 5 (5)
Pseudoaneurysm due to pancreatic fistula (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Intensive Care Unit or Progressive Care Unit Stay (General disorders) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SEAMGUARD With Bioabsorbable Staple (N=32) | TissueLink With Radiofrequency Ablation (N=35)
Pancreatic fistula drainage longer than 3 weeks (Gastrointestinal disorders) | 5 (5) | 9 (9)
Drained Amylase 3 Times Normal Upper Limit (Gastrointestinal disorders) | 15 (15) | 23 (23)
Specific Treatment for Pancreatic Fistula (Gastrointestinal disorders) | 4 (4) | 8 (8)
Pancreatic Fistula Documented by X-Ray (Gastrointestinal disorders) | 4 (4) | 5 (5)
Postoperative Infection (Infections and infestations) | 7 (7) | 8 (8)

LIMITATIONS AND CAVEATS:
The trial closed early due to poor accrual of subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No